CLINICAL TRIAL: NCT04465760
Title: A Phase II Study of Xisomab 3G3, a Monoclonal Antibody Preventing the Activation of FXI by FXIIa, for the Prophylaxis of Catheter-Associated Thrombosis
Brief Title: Xisomab 3G3 for the Prevention of Catheter-Associated Thrombosis in Patients With Cancer Receiving Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual rate
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Joseph Shatzel M.D., Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00018976; NCI-2020-02554 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00018976 (Other: OHSU Knight Cancer Institute); R01HL151367 (NIH)
Record Dates: First submitted 2020-06-25; First posted 2020-07-10 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Lymphoma; Malignant Solid Neoplasm; Plasma Cell Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — AB023

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive Care (xisomab 3G3) (Experimental): Patients receive xisomab 3G3 IV or via catheter within 48 hours of catheter placement. Patients then receive standard of care chemotherapy 2 days later. After approximately 2 weeks, patients undergo standard of care ultrasound for possible CAT.
  Interventions: Drug: Xisomab 3G3

INTERVENTIONS:
Drug: Xisomab 3G3 — Given IV or via catheter
  Other Names: AB 023; AB-023; AB023; Anti-factor XI Monoclonal Antibody Xisomab 3G3; Anti-FXI Antibody Xisomab 3G3

SUMMARY:
This phase II trial studies how well xisomab 3G3 works in preventing catheter-associated blood clots (thrombosis) in patients with cancer receiving chemotherapy. Many patients with cancer develop blood clots from their catheters and can have pain, swelling, and other symptoms. They also often require blood thinners, which can increase the risk of bleeding. Xisomab 3G3 is type of drug called a monoclonal antibody that may prevent blood clots caused by a catheter in patients receiving chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE I. To determine the efficacy of xisomab as measured by the incidence of catheter-associated thrombosis (CAT) in individuals with a central venous catheter.

SECONDARY OBJECTIVE:

I. To evaluate the safety and tolerability of xisomab 3G3 in cancer patients with a PICC or indwelling catheter.

EXPLORATORY OBJECTIVE:

I. Assessment of drug exposure and catheter occlusions leading to medical intervention.

OUTLINE:

Patients receive xisomab 3G3 intravenously (IV) or via catheter within 48 hours of catheter placement. Patients then receive standard of care chemotherapy 2 days later. After approximately 2 weeks, patients undergo standard of care ultrasound for possible CAT.

After completion of study, patients are followed up for 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Participant or legally authorized representative (LAR) must provide written informed consent before any study-specific procedures or interventions are performed
* In consultation with principal investigator (PI) and treating physician, participant's cancer-directed therapy allows for a 1-day period between administration of study drug and subsequent start of planned cancer-directed therapy
* Individuals with a confirmed solid malignancy that are scheduled to undergo insertion of a PICC line or indwelling central venous catheter as part of planned anticancer therapy per institutional standards
* Must have Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Platelet count > 100 x 10^9/L
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Participants of childbearing potential are defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and is not postmenopausal
* Female participants of childbearing potential must agree to use adequate methods of contraception starting with the first dose of study therapy through 90 days after the last dose of study therapy. Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year without an alternative medical cause
* Male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through 90 days after the last dose of study therapy

Exclusion Criteria:

* Actively receiving treatment in another therapeutic clinical trial
* Active acute leukemia (lymphoma and myeloma are allowed)
* At time of enrollment, known contraindication to anticoagulation therapy, including:

  * Clinically significant active bleeding
  * Individual is within 72 hours of major surgery
  * Abnormal baseline coagulation tests, including international normalized ratio (INR) > 1.5, or activated partial thromboplastin time (aPTT) prolonged
  * Abnormal renal function defined by an estimated glomerular filtration rate (eGFR) < 45 mL/min
  * Abnormal hepatic function defined as liver function tests (LFTs) (aspartate aminotransferase [AST], alanine aminotransferase [ALT] or total bilirubin) > 2 x the upper limit of normal or known Child-Pugh class B or C cirrhosis
  * Prior history of intracranial hemorrhage
  * Primary brain tumors or known brain metastasis
  * Major extracranial bleed within the last 6 months where the cause has not been identified or treated
  * Known bleeding diathesis
  * Use of therapeutic anticoagulation or anti-platelet agents for any indication at enrollment
  * At the discretion of the investigator, any other contraindication to anticoagulation therapy
  * Presence of a pediatric-sized PICC line
  * Participant is expected to receive chemotherapy associated with a 15% or higher incidence of grade 3-4 thrombocytopenia within 14 days of receiving study drug
* Preexisting intravenous catheter, or indwelling spinal or epidural catheter, at time of enrollment that is intended to remain for the duration of study. Participants may remain eligible if existing catheter is to be removed before placement of a catheter for cancer directed therapy. Removal of existing catheter should occur at least 24 hours prior to PICC or indwelling catheter insertion
* Previously documented hypersensitivity to either the drug or excipients
* Psychiatric illness/social situations, or any other condition, that in the opinion of the investigator, would limit compliance with study requirements
* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 90 days after the last dose of trial treatment
* Participant is allergic to heparin or heparin derivatives
* Participants with a history of venous thromboembolism within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Shatzel, M.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Derived] Pfeffer MA, Kohs TCL, Vu HH, Jordan KR, Wang JSH, Lorentz CU, Tucker EI, Puy C, Olson SR, DeLoughery TG, Hinds MT, Keshari RS, Gailani D, Lupu F, McCarty OJT, Shatzel JJ. Factor XI Inhibition for the Prevention of Catheter-Associated Thrombosis in Patients With Cancer Undergoing Central Line Placement: A Phase 2 Clinical Trial. Arterioscler Thromb Vasc Biol. 2024 Jan;44(1):290-299. doi: 10.1161/ATVBAHA.123.319692. Epub 2023 Nov 16. PMID 37970718

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care (Xisomab 3G3)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Xisomab 3G3)
Number analyzed (Participants) | 9
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 1
  40-49 years | 1
  50-59 years | 3
  60-69 years | 2
  70-79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Catheter-associated Thrombosis (CAT)
Description: The incidence of overall CAT (inclusive of both symptomatic and asymptomatic events) will be assessed and reported with 95% confidence interval.
Time Frame: Up to end of treatment visit (day 18)
Population: Eight of nine participants underwent screening ultrasound for catheter thrombosis. One patient had their catheter removed prior to screening ultrasound.
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Xisomab 3G3)
Number analyzed (Participants) | 8
Participants | 1

2. Secondary Outcome: Incidence of Major and Clinically-relevant Bleeding
Description: Bleeding will be defined using the International Society of Thrombosis and Hemostasis definition of major bleeding for clinical investigations of anti-hemostatic medicinal products in nonsurgical patients (i.e., fatal bleeding, critical organ bleeding such as central nervous system bleeding, or bleeding causing a fall in hemoglobin of 20 g/L or more) and clinically relevant non-major bleeding (i.e., bleeding that does not fit the former definition of major bleeding but prompts medical attention). The incidence of major and clinically relevant non-major bleeding, along with 95% confidence interval, will be assessed using the safety analysis set (all patients who are exposed to the single dose of study drug).
Time Frame: Up to end of follow-up (60 days from time of administration)
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Xisomab 3G3)
Number analyzed (Participants) | 9
Participants | 0

3. Secondary Outcome: Incidence of Xisomab 3G3-associated Adverse Events (AEs)
Description: Descriptive statistics of safety will be presented using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 using the safety analysis set (all patients who are exposed to the single dose of study drug). All on-study AEs, treatment-related AEs, serious adverse events (SAEs), and treatment-related SAEs will be tabulated using worst grade per National Cancer Institute (NCI) CTCAE v5.0 criteria by system organ class and preferred term. On-study lab parameters including hematology, chemistry, liver function, and renal function will be summarized using worst grade NCI CTCAE v5.0 criteria.
Time Frame: Up to end of follow-up (60 days from time of administration)
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Xisomab 3G3)
Number analyzed (Participants) | 9
Participants | 0

4. Other Pre Specified Outcome: Quantification of Coagulation Measures: Platelet Count
Description: Presented with descriptive statistics.
Time Frame: Up to end of treatment visit (day 18)
Measure: Mean (Standard Deviation); unit: cells*K/mm^3
Arm/Group | Supportive Care (Xisomab 3G3)
Number analyzed (Participants) | 9
cells*K/mm^3 | 275 (68)

5. Other Pre Specified Outcome: Quantification of Coagulation Measures: Prothrombin Time/International Normalized Ratio (PT/INR)
Description: Presented with descriptive statistics.
Time Frame: Up to end of treatment visit (day 18)
Measure: Mean (Standard Deviation); unit: INR
Arm/Group | Supportive Care (Xisomab 3G3)
Number analyzed (Participants) | 9
INR | 1.01 (0.01)

6. Other Pre Specified Outcome: Quantification of Coagulation Measures: Activated Partial Thromboplastin Time (aPTT)
Description: Presented with descriptive statistics.
Time Frame: Up to end of treatment visit (day 18)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Supportive Care (Xisomab 3G3)
Number analyzed (Participants) | 9
Seconds | 50.76 (2.81)

7. Other Pre Specified Outcome: Xisomab 3G3 Pharmacokinetics
Description: Presented with descriptive statistics.
Time Frame: Up to end of treatment visit (day 18)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Time to Detection of Thrombosis
Description: Will be reported for those (expected few) subjects with symptomatic CAT.
Time Frame: From xisomab 3G3 infusion up to end of treatment visit (day 18)
Population: No participants developed symptomatic CAT.
Arm/Group | Supportive Care (Xisomab 3G3)
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Time to Clot Symptoms
Description: Will be reported for those (expected few) subjects with symptomatic CAT.
Time Frame: From xisomab 3G3 infusion up to end of treatment visit (day 18)
Population: No participants developed symptomatic CAT.
Arm/Group | Supportive Care (Xisomab 3G3)
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Proportion of Patients That Had a Catheter Occlusion Requiring Medical Intervention
Description: Results will be presented with descriptive statistics.
Time Frame: Up to end of treatment visit (day 18)
Population: No participants developed catheter occlusion requiring medical intervention prior to the end of treatment visit.
Arm/Group | Supportive Care (Xisomab 3G3)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days post administration of the study drug.
Arm/Group | Supportive Care (Xisomab 3G3)
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Supportive Care (Xisomab 3G3) (N=9)
Mucositis oral (Gastrointestinal disorders) | 1
Vaginal yeast infection (Reproductive system and breast disorders) | 1
GI upset (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Access site pain (Skin and subcutaneous tissue disorders) | 1
Access site erythema (Skin and subcutaneous tissue disorders) | 1
Peripheral neuropathy (Nervous system disorders) | 2
Cold sensitivity (Nervous system disorders) | 5
Access site bruise (Skin and subcutaneous tissue disorders) | 1
Arm pain (Nervous system disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Gum bleeding (Gastrointestinal disorders) | 1
Epistaxis (Vascular disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Hypertension (Cardiac disorders) | 1
Rectal bleeding (Gastrointestinal disorders) | 1
Paresthesia (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 1
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Jaw pain (Nervous system disorders) | 1
Eye floaters (Eye disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Postoperative pain (Injury, poisoning and procedural complications) | 1
Non cardiac- chest pain (Nervous system disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Fatigue (General disorders) | 3
Loss of appetite (Metabolism and nutrition disorders) | 2
Lower extremity edema (General disorders) | 1
Shoulder pain (General disorders) | 1
Joint pain (General disorders) | 1
Body Ache (General disorders) | 1
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT04465760/Prot_SAP_000.pdf